CLINICAL TRIAL: NCT04816734
Title: Validation of an Educational Evaluation Plan and Assessment of Its Usefulness in Therapeutic Patient Education: Case of Pediatric Home Parenteral Nutrition
Brief Title: Initial Parenteral Nutrition Education of Parent Assessment Plan
Acronym: DISEPEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP200894; 2020-A01159-30 (Other: ID-RCB Number)
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Parenteral Nutrition
Keywords: Parenteral nutrition; Pediatric home parenteral nutrition; Parental therapeutic education; Educational evaluation
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parents (Experimental): Parents of children in need of home parenteral nutrition and participating in initial therapeutic education program of Necker-Enfants Malades hospital.
  Interventions: Other: Self-report questionnaires

INTERVENTIONS:
Other: Self-report questionnaires — Evaluation system of initial therapeutic education program about pediatric home parenteral nutrition.
  The assessment takes place after the parents have participated in the therapeutic education program and before their child returns home.

SUMMARY:
The department of gastroenterology, hepatology and pediatric nutrition at the Necker-Enfants Malades hospital has created an evaluation system for the initial therapeutic education program followed by parents of children requiring parenteral nutrition at the Necker-Enfants Malades hospital.

The aim of the study is to test this evaluation plan and assess its interest in the learning process of parents and then include it in the initial therapeutic education program for parents of children requiring parenteral nutrition of Necker-Enfants Malades hospital.

DETAILED DESCRIPTION:
Due to the highly technical nature of the care to be provided at home by parents of children in need of parenteral nutrition, an assessment of the acquisition of both factual knowledge provided to parents in hospital, but also of the reasoning, decision-making, technical skills and parents attitudes seem necessary and essential before the child's return to his home in order to guarantee his safety.

The department of gastroenterology, hepatology and pediatric nutrition of Necker-Enfants Malades hospital has developed an educational assessment system based on previous studies in this field. Composed of 4 tools, this plan allows a complete assessment with relevant educational decision fields of the set of skills that parents must master to cope with their child's illness on a daily basis, following their participation in the initial program of therapeutic education offered by the Necker hospital team.

The aim of the study is to test this evaluation plan and assess its interest in the learning process of parents and then include it in the initial therapeutic education program for parents of children requiring parenteral nutrition of Necker-Enfants Malades hospital.

ELIGIBILITY:
Inclusion Criteria:

* Holders of parental authority for children with parenteral nutrition participating in the initial education program of pediatric home parenteral nutrition of Necker hospital.
* informed consent signed by the patient and the investigator.
* patient affiliated to a social security scheme (beneficiary or beneficiary).

Exclusion Criteria:

* Subject having difficulty understanding the French language.
* Illiterate subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Usefulness by parent | Day 1
  Perceived usefulness of the evaluation session by the learners -parents- collected via a self-report questionnaire.
  4-point Likert scale: Strongly agree, Somewhat agree, Somewhat disagree, Disagree.

SECONDARY OUTCOMES:
Usefulness by carer | Day 1
  Perceived usefulness of the evaluation session by users -carers- collected via a self-report questionnaire.
  4-point Likert scale: Strongly agree, Somewhat agree, Somewhat disagree, Disagree.
Educational quality by parent | Day 1
  Educational quality of the 4 assessment tools, assessed via 4 self-report questionnaires intended for parents.
  4-point Likert scale: Strongly agree, Somewhat agree, Somewhat disagree, Disagree.
Educational quality by carer | Day 1
  Educational quality of the 4 assessment tools, assessed via 4 self-report questionnaires intended for carers.
  4-point Likert scale: Strongly agree, Somewhat agree, Somewhat disagree, Disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile LAMBE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Cécile GODOT, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No